CLINICAL TRIAL: NCT02843867
Title: Influence de l'ORientation de la réponse LYmphocytaire Sur la Survenue de Complications athéromateuses après Transplantation rénale (étude ORLY-EST 2)
Brief Title: Orientation of the Lymphocyte Response to the Occurrence of Atherosclerotic Complications After Kidney Transplantation
Acronym: ORLY-Est
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University of Franche-Comté (Other); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Other Study IDs: R/2011/44
Record Dates: First submitted 2016-07-08; First posted 2016-07-26 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Transplantation; Immunology; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Peripheral Blood Mononuclear Cells
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood sample — 36 ml of blood sample at D0 and 1 year after transplantation

SUMMARY:
The incidence of atherosclerotic complications is increased after kidney transplantation. Traditional risk factors do not fully explain this increased risk. Atherosclerosis is an inflammatory disease in which all players in the immune response are involved. The impact of these immune responses is not well known in immunocompromised patients, particularly among organ transplant. Nevertheless, the work of our group suggest that innate and acquired responses through different mechanisms influencing the evolution of atheromatous disease after transplantation.

The investigators therefore propose to study the impact of the expansion of regulatory T cells on the risk of atherosclerotic complications after transplantation.

Since November 2008, the investigators began a multicenter, prospective study whose purpose is to study in detail the immunological mechanisms of atherosclerosis after transplantation via immunomonitoring cohort of renal transplant patients in the Grand East Interregion. It was planned to include 500 patients and to date a little more than half have been included. After completion of the blood test, the tubes are routed over the Biomonitoring Platform (CIC-BT 506 Besançon) and the samples are stored in CRB Dijon.

The atherosclerotic events are recorded prospectively. The investigators hope to implement as part of ORLY IS, a second study to determine the impact of an expansion of regulatory T cells on the risk of atherosclerotic events.

Our hypothesis is that a cell rate regulatory T below the median results in an increase of 5% of atherosclerotic complications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged over 18 years
2. Patients receiving a renal transplant
3. Patients able to understand the benefits and risks of testing
4. Patients gave written informed consent.

Exclusion Criteria:

1. Inability to understand the advantages and disadvantages of the study; psychiatric disorders judged by the investigator to be incompatible with the inclusion in the study.
2. Immunosuppressive therapy immediately prior to transplantation
3. Cancer (except skin cancer) or malignant blood disease being treated; active infection; decompensated cirrhosis [patients had cancer and considered as cured or in remission, patients with virus infection of hepatitis B or hepatitis C and having no cirrhosis may be included].

This study is strictly non-interventional, participation in another study is not a cons-indication to the inclusion in this study and no exclusion period is required for inclusion in another study after inclusion in this study (Art L. 1121-12 (loi n°2004-806 du 9 Août 2004).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to 1000 patients receiving a renal transplant in Hospital of Besançon, Dijon, Nancy, Reims, Clermont-Ferrand, Strasbourg et Kremlin-Bicêtre.
Sampling Method: Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2008-11-28 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2030-10-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of regulatory T cells related to atherosclerotic complications events. | 5 or 10 years
  Percentage of regulatory T cells

SECONDARY OUTCOMES:
Atherosclerotic complications events | 5 or 10 years
  Percentage of regulatory T cells
Genetic determinants (TNF-alpha, IL-6,...) related to cardiovascular events | 5 or 10 years
  Percentage of regulatory T cells

CONTACTS AND LOCATIONS:
Overall Officials: Didier Ducloux, Pr., Principal Investigator — CHRU de Besançon
Locations (7):
- France (7):
  - CHU de Besançon, Besançon
  - CHU Clermont-Ferrand, 58 rue Montalembert, 63003 Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Hôpital du Bocage, 2 Bd du Maréchal de Lattre de Tassigny, 21079 Dijon cedex, Dijon
  - Hôpital du Kremlin Bicêtre 78, rue du Général Leclerc, 94275 Le Kremlin-Bicêtre Cedex, Le Kremlin-Bicêtre
  - CHU Brabois, et Vandoeuvre les Nancy, Nancy
  - CHU Reims, 45 rue Cognacq-Jay 51092 Reims Cedex, Reims
  - Hôpital Civil- 1, place de l'hôpital BP426 ; 67091 Strasbourg Cedex, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
Identified individual participant data for all outcome measures will be made available within 6 monts of study completion

REFERENCES:
- [Derived] Ducloux D, Courivaud C, Bamoulid J, Crepin T, Gaiffe E, Laheurte C, Vauchy C, Rebibou JM, Saas P, Borot S. Immune phenotype predicts new onset diabetes after kidney transplantation. Hum Immunol. 2019 Nov;80(11):937-942. doi: 10.1016/j.humimm.2019.08.006. Epub 2019 Sep 10. PMID 31515130
- [Derived] Ducloux D, Legendre M, Bamoulid J, Rebibou JM, Saas P, Courivaud C, Crepin T. ESRD-associated immune phenotype depends on dialysis modality and iron status: clinical implications. Immun Ageing. 2018 Jul 17;15:16. doi: 10.1186/s12979-018-0121-z. eCollection 2018. PMID 30026783